CLINICAL TRIAL: NCT07406412
Title: HoCa - A Multidimensional Study on Menopausal Hormonal Change, Cardiometabolic Health and Embodied Experience
Brief Title: Hormonal Regulation of Cardiometabolic Health Study
Acronym: HoCa
Status: Not yet recruiting | Type: Observational
Sponsor: University of Jyvaskyla (Other)
Collaborators: Wellbeing Services County of Central Finland (Unknown); Wellbeing Services County of North Savo (Unknown); Wellbeing Services County of Pirkanmaa (Other); Wellbeing Services County of Southwest Finland (Unknown); Wellbeing Services County of North Ostrobothnia (Unknown); Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Sponsor
Other Study IDs: 2U/2025/HoCa
Record Dates: First submitted 2026-01-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Menopause Surgical
Keywords: Oophorectomy; Menopause; Estrogen Deficiency; Cardiometabolic Health; Quality of Life; Body Composition; Physical performance; Neurophysiology; Prospective observational study; Embodied experience; Health behavior; Adipose Tissue; Fat Oxidation; Vascular function; Menopause symptoms
MeSH Terms: conditions — Health Behavior | interventions — Ovariectomy; Hormone Replacement Therapy; mahuang-tang

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected for leukocyte and platelet analyses, including flow cytometry and transcriptomic profiling (microRNA and mRNA). Plasma and serum samples will be retained for biomarker assays related to hormonal, metabolic, and inflammatory status. Samples will be obtained at rest and after a standardised cycle ergometer test to assess exercise-induced responses. In addition, subcutaneous and visceral adipose tissue samples collected during oophorectomy will be used for organoid-based studies of adipose tissue health and cellular function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Menopause Cohort: Women aged 35-50 undergoing bilateral (or unilateral, if one ovary remains) oophorectomy for non-malignant indications.
  Interventions: Procedure: Surgical removal of ovaries; Drug: Hormone Replacement Therapy (HRT)

INTERVENTIONS:
Procedure: Surgical removal of ovaries — Bilateral oophorectomy, or unilateral if only one ovary remains. Other organs may also be removed during the same procedure, such as fallopian tubes (salpingectomy) and/or uterus (hysterectomy).
  Other Names: oophorectomy
Drug: Hormone Replacement Therapy (HRT) — Post-surgery HRT as part of clinical treatment after the 1-2 month follow-up. HRT may be any commercially available systemic treatment.
  Other Names: systemic menopausal hormone therapy; MHT

SUMMARY:
The goal of this observational study is to understand how the loss of ovarian function after oophorectomy affects the health and well being of women aged 35-50.

The study focuses on four areas:

1. Quality of life and embodied experience,
2. Cardiometabolic health,
3. Central nervous system function, and
4. Adipose tissue health and cellular function.

Our primary goal is to understand the effects of oophorectomy on women's health in focus areas 1 to 3. To do this, we will compare women's health before surgery with follow up assessments at 1-2 months and 12 months after surgery. Some participants may start hormone replacement therapy (HRT) during follow up as part of their routine care; this is outside the study protocol. As an exploratory aim, we will examine whether 12 month outcomes-or the change from baseline to 12 months-differ between participants who begin HRT and those who do not.

Focus area 4 provides an opportunity to explore how molecular and cellular mechanisms in adipose tissue respond to the loss of ovarian hormones. These analyses are exploratory and intended to offer mechanistic insight rather than clinical endpoints.

Participants will:

* undergo bilateral (or unilateral, if only one ovary remains) oophorectomy as part of their clinical treatment,
* complete questionnaires and physiological measurements at three time points,
* a subgroup will participate in qualitative interviews about their lived experience of surgical menopause,
* and a subgroup will volunteer adipose tissue samples collected during surgery.

DETAILED DESCRIPTION:
Overview

This observational longitudinal study investigates how the abrupt loss of ovarian function following bilateral (or unilateral, if only one ovary remains) oophorectomy affects the health and well being of women aged 35-50 years. Surgical menopause induces rapid endocrine, metabolic, vascular, neural, and psychosocial changes. To capture these adaptations comprehensively, the study evaluates four interconnected domains: (1) quality of life and embodied experience, (2) cardiometabolic health, (3) central nervous system function, and (4) adipose tissue health and cellular function.

Participants undergo assessments at three time points: pre surgery, 1-2 months post surgery, and 12 months post surgery. These visits include validated questionnaires, physiological and neuromuscular tests, vascular and exercise assessments, and the collection of blood samples at rest and after a standardised cycle ergometer test. A subgroup participates in qualitative interviews at all visits, and another subgroup donates adipose tissue samples during surgery for exploratory cellular analyses.

Some participants may begin hormone replacement therapy (HRT) after the 1-2 month visit as part of their clinical care. Because HRT initiation is outside the study protocol, HRT related comparisons (e.g., whether 12 month outcomes or change from baseline differ between HRT starters and non starters) will be conducted exploratorily, following definitions and modelling approaches described in the Statistical Analysis Plan.

Blood samples are analysed for a broad panel of metabolic, inflammatory, hormonal, and exercise responsive biomarkers to characterise systemic adaptations to surgical menopause. These biomarker analyses are exploratory and intended to provide mechanistic insight; they are not registered as outcome measures.

This four domain structure enables the study to integrate patient reported outcomes, whole body physiology, neural activation, vascular regulation, exercise metabolism, and adipose tissue biology, offering a multidimensional understanding of how surgical menopause impacts women's health over time.

Domain 1: Quality of Life and Embodied Experience

Surgical menopause can cause a variety of symptoms and affect daily functioning, health behaviours, and overall quality of life. We collect patient-reported outcomes using validated questionnaires covering quality of life, menopausal symptoms, sleep, pelvic floor symptoms, sexual function, psychosocial dimensions, and health behaviours such as physical activity and eating patterns. Participants also complete a food diary and wear a 7-day accelerometer to provide objective measures of dietary intake and physical activity. In addition, a subgroup participates in qualitative interviews, which help deepen our understanding of the lived experience of surgical menopause.

Primary outcomes in this domain are the RAND-36 total score and the Menopause Rating Scale (MRS) total score, which capture changes in broad health-related quality of life and menopausal symptom burden following oophorectomy.

Secondary outcomes include the Women's Health Questionnaire (WHQ), Pelvic Floor Distress Inventory-20 (PFDI-20), and the Athens Insomnia Scale-5 (AIS-5), providing a more detailed understanding of psychosocial health, pelvic floor symptoms, and sleep quality.

Other prespecified outcomes contribute additional context on general well-being, emotional functioning, health behaviours, and embodied experiences. These include the 15D, Female Sexual Function Index (FSFI), Center for Epidemiological Studies Depression Scale (CES-D), Satisfaction With Life Scale (SWLS), Positive and Negative Affect Schedule (PANAS), Eating Disorder Examination Questionnaire (EDE-Q), Three-Factor Eating Questionnaire-R18 (TFEQ-R18), the International Physical Activity Questionnaire-Short Form (IPAQ-SF), and a 4-item Finnish physical activity questionnaire. These measures extend the scope of quality-of-life assessment and support interpretation of primary and secondary outcomes.

Finally, qualitative interviews conducted with a subgroup of participants at each time point provide rich insights into bodily changes, identity, emotions, and the lived experience of surgical menopause. These interviews enhance the interpretation of questionnaire-based findings and allow a more integrated understanding of women's experiences during the transition to surgical menopause.

Domain 2: Cardiometabolic Health

Loss of ovarian function following oophorectomy may influence whole-body metabolism, body composition, vascular regulation, and exercise capacity. To characterise these possible adaptations, cardiometabolic health is assessed at each visit with standardized protocols that include indirect calorimetry, body composition measurements, vascular assessments, and exercise physiology testing using standardised cycle ergometer tests. Together, these measures help us evaluate whether endocrine changes are associated with alterations in metabolic rate, adiposity, cardiovascular function, and exercise-related responses over time.

Primary outcomes in this domain are resting energy expenditure (REE), total fat mass (FM), and aortic pulse wave velocity (PWV). These endpoints capture core aspects of metabolic function, whole body adiposity, and arterial stiffness-parameters that may change after the loss of ovarian function and are relevant to longer-term cardiometabolic risk.

Secondary outcomes include fat-free mass (FFM), augmentation index (AIx) as an additional marker of arterial wave reflection, and peak fat oxidation during exercise, offering insight into potential shifts in metabolic flexibility and substrate use at submaximal workloads.

Other prespecified outcomes provide supporting information on anthropometry, muscular performance, vascular regulation, and exercise responses. These include body mass index (BMI), waist circumference, handgrip strength, knee extension strength, and countermovement jump (CMJ) height. Additional central hemodynamic measures-aortic systolic and diastolic blood pressure, aortic pulse pressure, and reflection time-further characterise vascular load.

Microvascular and tissue-level parameters include forearm Laser Doppler readings (baseline perfusion, endothelium-dependent vasodilation, post-occlusive reactive hyperemia) and quadriceps near-infrared spectroscopy (NIRS) measures (resting StO2, minimum StO2 during exercise, StO2 recovery slope, total hemoglobin). Exercise metabolism is additionally profiled using peak oxygen uptake (VO2peak), resting fat oxidation rate, and maximal fat oxidation rate (MFO).

Exploratory blood biomarkers (not registered as outcomes) At each visit, venous blood samples are collected at rest and after the standardised cycle ergometer test. These samples will be analysed for exploratory biomarkers, including a broad panel of metabolic, inflammatory, and hormonal markers, to characterise systemic adaptations to the loss of ovarian function after oophorectomy and to examine potential changes in exercise responses. These biomarker analyses are exploratory and intended to provide mechanistic insight; they are not registered as outcome measures and follow definitions and procedures described in the Statistical Analysis Plan.

Domain 3: Central Nervous System Function

Loss of ovarian function following oophorectomy may influence neural activation, neuromuscular performance, and corticospinal and reticulospinal responsiveness. To characterise these possible adaptations, a subsample of participants completes a set of standardised neurophysiological assessments, including isometric strength testing, reaction time tasks, and transcranial magnetic stimulation (TMS). These tests provide complementary insight into neural drive to muscle and the excitability of corticospinal and cortico reticulospinal pathways during the first postoperative year.

No primary outcomes are defined for this domain. Secondary outcomes in this domain quantify neural activation and corticospinal responsiveness using complementary physiological measures. Maximum isometric voluntary contraction force (MVC) is assessed to evaluate volitional muscle activation during isometric elbow flexion. A StartReact test assesses reaction time and the StartReact effect, defined as the difference in reaction time between quiet and loud sound conditions. Cortical excitability is assessed using single pulse TMS, with the main analysis variable being motor evoked potential (MEP) amplitude normalised to the maximal compound muscle action potential (Mmax), elicited via peripheral nerve stimulation.

Other prespecified outcomes further characterise neuromuscular and corticospinal function. Rate of torque development (RTD) and voluntary electromyography (EMG) amplitude (0-50 ms) are derived from force and EMG signals recorded during the StartReact test. Paired pulse TMS methods are used to quantify short interval intracortical inhibition (SICI), long interval intracortical inhibition (LICI), and intracortical facilitation (ICF) relative to single pulse comparator responses. StartleTMS, which pairs a loud acoustic stimulus with TMS, provides an additional measure of startle related facilitation of corticospinal output. Silent period duration is measured during single pulse TMS and then normalised to MEP amplitude to enable comparison across time points.

Together, these measures provide a multidimensional characterisation of neural responsiveness, including voluntary activation, intracortical inhibitory and facilitatory circuits, and the excitability of corticospinal and cortico reticulospinal pathways.

DOMAIN 4: Adipose Tissue Health and Cellular Function

Loss of ovarian function following oophorectomy may be associated with changes in adipose tissue biology, including cellular composition, lipid handling, inflammatory signalling, and gene expression. To explore these potential mechanisms, a subsample of participants donates subcutaneous and, where available, visceral adipose tissue during surgery. From these tissues, adipose organoids ("Adipoids") are developed and exposed to controlled hormonal environments (e.g., defined hormones or conditioned media supplemented with pre and postmenopausal sera) to model post oophorectomy conditions in vitro.

This domain is considered exploratory; thus, no primary or secondary outcomes are described. We describe one other prespecified outcome (exploratory mechanistic readout): Hormonal Regulation of Adipose Tissue Health and Cellular Function, which refers to a change in Adipoid cellular content/cellularity (e.g., nuclei count or cells/mL) in response to a change in hormonal environment. We will also perform additional mechanistic assays (exploratory; not registered as outcome measures), including

* Lipid uptake/handling
* Responses to inflammatory stimuli
* Gene expression profiles
* Secretome characteristics

These laboratory analyses aim to reveal molecular pathways through which the loss of ovarian hormones may affect adipose biology. They are exploratory, not intended as clinical endpoints, and follow laboratory Standard Operation Protocols and the Statistical Analysis Plan.

Exploratory analyses of Hormone Replacement Therapy (HRT)

Some participants may begin hormone replacement therapy (HRT) after the 1-2 month visit as part of their routine clinical care. Because HRT initiation is outside the study protocol, comparisons involving HRT are conducted exploratorily. These analyses examine whether 12 month outcomes-or the change from baseline to 12 months-differ between HRT starters and non starters. HRT exposure will be defined using time varying information collected at each visit, and sensitivity analyses will explore alternative exposure windows. All analytic approaches, including covariate selection and handling of missing data, are prespecified in the Statistical Analysis Plan. These exploratory analyses do not constitute registered outcome measures for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-50 years
* Pre- or perimenopausal status (defined as self-reported menstrual bleedings and/or follicle-stimulating hormone ≤25 IU/L)
* One or two functional ovaries
* Planning to undergo bilateral oophorectomy or salpingo-oophorectomy (BSO) or unilateral oophorectomy or salpingo-oophorectomy (SO) if the other ovary has been previously removed, for non-malignant reasons

Exclusion Criteria:

* Oophorectomy due to ovarian cancer or other malignant conditions
* Current systemic estrogen-containing medication

The following exclusion criteria apply only to participation in physiological assessments (not questionnaires or interviews):

* Severe heart or liver disease
* Mobility limitations that prevent participation in physical exercise tests

The following factors do not lead to exclusion but will be recorded and considered in analyses:

* Use of medications such as weight reduction drugs, lipid-lowering agents, or antihypertensives
* Concomitant hysterectomy or other surgeries performed with oophorectomy
* Use of local vaginal oestrogen therapy
* Initiation of systemic hormone replacement therapy (HRT) after the 1-2-month post-surgery assessments (allowed according to clinical need; not part of the study protocol)

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from gynaecological surgical waiting lists at the university and central hospitals across Finland. Recruitment sites include the Wellbeing Service counties of Central Finland, North Savo, Pirkanmaa, Southwest Finland, and North Ostrobothnia, as well as the Hospital District of Helsinki and Uusimaa (HUS).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in RAND-36 Item Health Survey (RAND-36) Total Score | Baseline to 1-2 months and 12 months post-surgery
  The RAND-36 Item Health Survey is a 36-item health-related quality of life instrument with eight domains: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health, Vitality, Social Functioning, Role Limitations due to Emotional Problems, and Emotional Well-Being. Each domain is scored on a 0-100 scale; higher scores indicate better health status. The RAND-36 total score is computed as the arithmetic mean of the eight domain scores (range 0-100; higher = better). The reported measure is the change from baseline to follow-up (follow-up minus baseline); positive values indicate improvement. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis may use a reduced/composite RAND-36 score (e.g., a domain subset with documented performance advantages); details are specified in the SAP. This sensitivity analysis is supportive and does not replace the prespecified analysis of this primary outcome.
Change from Baseline in Menopause Rating Scale (MRS) Score | Baseline to 1-2 months and 12 months post-surgery
  The Menopause Rating Scale (MRS) is an 11-item questionnaire assessing menopausal symptom burden across three domains: Somatic (4 items), Psychological (4 items), and Urogenital (3 items). Each item is scored 0-4 (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe), yielding a total score range of 0-44, where higher scores indicate worse symptom severity/health-related quality of life. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate worsening and negative values indicate improvement. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis may use a reduced MRS score that excludes items with documented suboptimal performance; details are specified in the Statistical Analysis Plan. This sensitivity analysis is supportive and does not replace the prespecified analysis of this primary outcome.
Change from Baseline in Resting Energy Expenditure (REE, kcal/day) Measured by Indirect Calorimetry | Baseline to 1-2 months and 12 months post-surgery
  Resting energy expenditure (REE) is measured by indirect calorimetry (ventilated hood; overnight fast 10-12 h; supine, thermoneutral room). After stabilization, VO2 and VCO2 are recorded for ≥20-30 min; a steady-state segment (e.g., ≥5 min with CV <10% and physiologic RQ) is used to compute REE (kcal/day) via the Weir equation, higher values = higher energy expenditure. Outcome is change from baseline to follow-up (follow-up - baseline); higher positive values = higher increase in energy expenditure. Procedures/quality criteria follow the device manual and the Statistical Analysis Plan (SAP). Per SAP, supportive analyses may adjust for body composition (FFM/FM) or express REE relative to FFM; these do not replace the prespecified analysis of this primary outcome.
Change from Baseline in Total Fat Mass (kg) Measured by Bioelectrical Impedance Analysis | Baseline to 1-2 months and 12 months post-surgery
  Total fat mass (FM) will be measured by bioelectrical impedance analysis (BIA; InBody) under standardized conditions, including a 10-12 h fast before assessment. FM is reported in kg; higher values indicate higher fat mass. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement procedures, quality criteria, and handling of missing/outliers follow the device manual and the Statistical Analysis Plan (SAP). Per SAP, a prespecified sensitivity analysis will estimate FM using DXA (where available); this analysis is supportive and does not replace the prespecified analysis of this primary outcome.
Change from Baseline in Aortic Pulse Wave Velocity (PWV, m/s) | Baseline to 1-2 months and 12 months post-surgery
  Aortic pulse wave velocity (PWV) will be measured using an oscillometric Arteriograph device under standardized resting conditions, including a 10-12 h fast and avoidance of vigorous physical activity during the previous 24 h. Measurements are taken supine in a quiet, thermoneutral room. PWV is reported in m/s; higher values indicate greater arterial stiffness. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures, calibration, and quality criteria follow the device manual and the Statistical Analysis Plan (SAP). Per SAP, supportive analyses may examine additional Arteriograph variables (e.g., AIx, aortic pressures); these do not replace the prespecified analysis of this primary outcome.

SECONDARY OUTCOMES:
Change from Baseline in Women's Health Questionnaire (WHQ) Total Score (36-item) | Baseline to 1-2 months and 12 months post-surgery
  The Women's Health Questionnaire (WHQ) is a 36-item instrument assessing midlife women's emotional and physical health across multiple domains (e.g., depressed mood, somatic symptoms, vasomotor symptoms, anxiety/fears, sleep problems, menstrual symptoms, sexual functioning, and memory/concentration). Domain scores are transformed to a 0-100 scale and averaged to a total score (range 0-100), where higher scores indicate worse health-related quality of life. The reported measure is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate worsening. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis may use a reduced WHQ total score that excludes items with documented suboptimal performance; details are specified in the SAP. This sensitivity analysis will not replace the prespecified analysis of this secondary outcome and will be interpreted as supportive.
Change from baseline in the Pelvic Floor Distress Inventory-20 (PFDI-20) total score (20-item) | Baseline to 1-2 months and 12 months post-surgery
  The Pelvic Floor Distress Inventory-20 (PFDI-20) is a 20-item questionnaire assessing pelvic floor symptom distress across three subscales: POPDI-6 (pelvic organ prolapse distress), CRADI-8 (colorectal-anal distress), and UDI-6 (urinary distress). Each subscale is scored 0-100, and the PFDI-20 total score is their sum (range 0-300), where higher scores indicate worse symptom distress and poorer health-related quality of life. The outcome is the change from baseline to the specified follow-up (follow-up minus baseline); positive values indicate worsening. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis will examine the three PFDI-20 subscale scores (POPDI-6, CRADI-8, UDI-6), each scored 0-100 (higher = worse). These analyses are supportive only and do not replace the prespecified analysis of the PFDI-20 total score as a secondary outcome.
Change from Baseline in Athens Insomnia Scale-5 (AIS-5) Score | Baseline to 1-2 months and 12 months post-surgery
  The Athens Insomnia Scale-5 (AIS-5) is a 5-item validated instrument assessing sleep difficulty. Each item is scored 0-3, producing a total score of 0-15, where higher scores indicate more severe insomnia symptoms. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate worsening. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis may examine individual AIS-5 items; these analyses are supportive only and do not replace the prespecified analysis of this secondary outcome.
Change from Baseline in Fat-Free Mass (kg) Measured by Bioelectrical Impedance Analysis | Baseline to 1-2 months and 12 months post-surgery
  Fat-free mass (FFM) will be measured by bioelectrical impedance analysis (BIA; InBody) under standardized conditions, including a 10-12 h fast before assessment. FFM is reported in kg; higher values indicate higher fat-free mass. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement procedures, quality criteria, and handling of missing/outliers follow the device manual and the Statistical Analysis Plan (SAP). Per SAP, a prespecified sensitivity analysis will estimate FFM using DXA (where available); this analysis is supportive and does not replace the prespecified analysis of this secondary outcome.
Change from Baseline in Augmentation Index (AIx, %) | Baseline to 1-2 months and 12 months post-surgery
  Augmentation Index (AIx) will be measured using the Arteriograph under the same standardized resting conditions, including a 10-12 h fast and avoidance of vigorous physical activity during the preceding 24 h. AIx is expressed in %; higher values indicate greater arterial wave reflection. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline). Measurement procedures and quality criteria follow the device manual and the Statistical Analysis Plan.
Change from Baseline in Peak Fat Oxidation During Exercise (g/min) | Baseline to 1-2 months and 12 months post-surgery
  During steady-state cycling at 45-50% of the peak power derived from the VO2peak test, whole-body fat oxidation will be measured by indirect calorimetry. The peak value during the bout will be recorded in g/min; higher values indicate higher fat oxidation during exercise. Pre-test conditions: 10-12 h fast and no vigorous physical activity in the prior 24 h. Outcome is change from baseline. Exercise protocol, data smoothing and calculation details follow the Statistical Analysis Plan.
Change from Baseline in Maximum Isometric Voluntary Contraction Force (MVC) [Newton, N] | Time Frame: Baseline to 1-2 months and 12 months post-surgery
  Testing is performed under controlled pre-test conditions (10-12 h fast, no vigorous physical activity in the prior 24 h), seated in a thermoneutral room. The participant performs 3-5 isometric elbow flexion actions by maximally contracting the biceps brachii muscle while seated in an electromechanical dynamometer. Force and electromyography (EMG) activity are recorded during the contractions. The outcome is the change in force (N) from baseline to the specified follow-up (follow-up - baseline). Condition, quality criteria, and analysis are defined in the Statistical Analysis Plan.
Change from Baseline in StartReact Effect (ms) [difference in reaction time between loud and quiet sound conditions] | Baseline to 1-2 months and 12 months post-surgery
  Reaction time, defined as the delay between the visual stimulus presentation and the increase in voluntary electromyography (EMG) signal amplitude above baseline (+7SD), is obtained through the StartReact test. Testing is performed under controlled pre-test conditions (10-12 h fast, no vigorous physical activity in the prior 24 h), seated in a thermoneutral room. The StartReact effect is reported in milliseconds (ms) as the difference in reaction time between quiet and loud sound conditions; higher values indicate a larger effect. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). In addition, the StartReact test provides data on rate of torque development (0-50 ms) and voluntary EMG amplitude (0-50 ms) as force and EMG are sampled simultaneously. These variables are collected but analyzed and reported separately as Other Prespecified Outcome Measures. Condition, quality criteria, and analysis are defined in the Statistical Analysis Plan.
Change from Baseline in Motor Evoked Potential (MEP) Amplitude (mV/Mmax) Measured by Transcranial Magnetic Stimulation | Baseline to 1-2 months and 12 months post-surgery
  Cortical excitability will be evaluated using transcranial magnetic stimulation (TMS) over the motor cortex with electromyography (EMG) recordings from the biceps during a light, standardised voluntary contraction. Pre-test conditions: 10-12 h fast and no vigorous physical activity in the prior 24 h; testing in a quiet, thermoneutral room with consistent coil positioning. The main analysis variable for this outcome is normalized MEP amplitude (mV/Mmax) throughout the stimulus-response curve; higher values indicate greater corticospinal responsiveness. Maximal compound muscle action potential (Mmax) is elicited by peripheral nerve stimulation and recorded from the same muscle using the same electrode configuration. The outcome is the change from baseline to follow up (follow up - baseline). Hot spot identification, motor thresholding, trial number/rejection rules, and averaging procedures follow the Statistical Analysis Plan.

OTHER OUTCOMES:
Change from Baseline in 15D Health-Related Quality of Life (15D) Index Score | Baseline to 1-2 months and 12 months post-surgery
  The 15D is a 15-dimension health-related quality of life instrument that yields a single index score ranging from 0 to 1, where higher scores indicate better health status. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate improvement. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). This measure is prespecified as Other Prespecified Outcome and will be interpreted as supportive.
Change from Baseline in Female Sexual Function Index (FSFI) Total Score | Baseline to 1-2 months and 12 months post-surgery
  The Female Sexual Function Index (FSFI) is a 19-item instrument covering six domains of sexual function (Desire, Arousal, Lubrication, Orgasm, Satisfaction, Pain). The FSFI total score ranges from 2 to 36, where higher scores indicate better sexual function. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate improvement. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). A prespecified sensitivity analysis may examine domain scores; these analyses are supportive only and do not replace the prespecified analysis of this outcome.
Change from Baseline in Center for Epidemiological Studies Depression Scale (CES-D) Total Score | Baseline to 1-2 months and 12 months post-surgery
  The CES-D consists of 20 items, each scored 0-3; the total score ranges from 0 to 60, where higher scores indicate greater depressive symptom severity. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate worsening. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). This measure is listed as an Other Prespecified Outcome and will be interpreted as supportive.
Change from Baseline in Satisfaction With Life Scale (SWLS) Score | Baseline to 1-2 months and 12 months post-surgery
  The SWLS has 5 items scored 1-7; total score 5-35, where higher scores indicate greater life satisfaction. Outcome is change from baseline to the specified follow-up (follow-up minus baseline); positive = improvement. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). Listed as Other Prespecified Outcome (supportive).
Change from Baseline in Positive Affect and Negative Affect Scores (PANAS) Total Scores | Baseline to 1-2 months and 12 months post-surgery
  The PANAS comprises two 10-item scales scored 1-5 each; Positive Affect and Negative Affect totals each range 10-50. Higher Positive Affect = better, higher Negative Affect = worse. Outcome is change from baseline to the specified follow-up (follow-up minus baseline); direction interpreted per subscale. Scoring follows the instrument manual and the Statistical Analysis Plan (SAP). Listed as Other Prespecified Outcomes (supportive).
Change from Baseline in Eating Disorder Examination Questionnaire (EDE-Q) Global Score | Baseline to 1-2 months and 12 months post-surgery
  The EDE-Q assesses eating-disorder psychopathology; the global score is the mean of four subscales, ranging 0-6, where higher scores indicate more severe pathology. Outcome is change from baseline to the specified follow-up (follow-up minus baseline); positive = worsening. Scoring follows the instrument manual and the Statistical Analysis Plan. Listed as Other Prespecified Outcome (supportive analysis).
Change from Baseline in Three-Factor Eating Questionnaire-R18 (TFEQ-R18) Subscale Scores | Baseline to 1-2 months and 12 months post-surgery
  The Three-Factor Eating Questionnaire-R18 (TFEQ-R18) assesses eating-related traits across three subscales: Cognitive Restraint (6 items), Uncontrolled Eating (9 items), and Emotional Eating (3 items). Items are scored 1-4 and each subscale score is the mean of its items linearly transformed to a 0-100 scale using (mean - 1) × 100 / 3; higher scores indicate more of the trait (i.e., greater restraint, greater uncontrolled eating, or greater emotional eating). Outcomes are the changes from baseline to the specified follow-up time point(s) (follow-up - baseline); direction is interpreted per subscale (e.g., higher Uncontrolled/Emotional Eating = worse, higher Cognitive Restraint = greater restraint; clinical desirability depends on context and is prespecified in the Statistical Analysis Plan [SAP]). Scoring and handling of missing items follow the instrument manual and the SAP.
Change from Baseline in the International Physical Activity Questionnaire-Short Form (IPAQ-SF) total amount of Physical Activity [MET-minutes/week] | Baseline to 1-2 months and 12 months post-surgery
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) provides a summary estimate of weekly physical activity expressed as MET-minutes/week, combining walking, moderate, and vigorous physical activities. Higher values indicate higher total physical activity. The outcome is the change from baseline to the specified follow-up (follow-up minus baseline). Scoring follows IPAQ guidelines and the Statistical Analysis Plan (SAP). This measure is listed as an Other Prespecified Outcome and will be interpreted as supportive.
Change from Baseline in Physical Activity (MET-hours/week) Assessed by the 4-Item Self-Reported Physical Activity Questionnaire | Baseline to 1-2 months and 12 months post-surgery
  The Self-Reported Physical Activity Questionnaire (Kujala et al., 1988) is a 4-item instrument assessing habitual weekly physical activity, including frequency, average duration, and typical intensity of leisure-time exercise. Responses are converted to MET-hours/week using standardized intensity estimates; higher values indicate higher physical activity. The outcome is the change from baseline to the specified follow-up time point (follow-up minus baseline); positive values indicate increased activity. Scoring and MET conversion follow the Statistical Analysis Plan (SAP). This measure is listed as an Other Prespecified Outcome and will be interpreted as supportive.
Qualitative Assessment of the Lived Experience of Surgical Menopause | Baseline, 1-2 months, and 12 months post-surgery
  Semi-structured interviews exploring participants' embodied perceptions and experiences of surgical menopause. Data will be analysed using qualitative thematic analysis to provide a contextual understanding of physiological findings.
Change from Baseline in Body Mass Index (BMI, kg/m²) | Baseline, 1-2 months, and 12 months post-surgery
  BMI is calculated as weight (kg) divided by height squared (m²). Weight is measured under standardized conditions at baseline and follow-ups; height is measured at baseline only. BMI is expressed as kg/m²; higher values indicate higher body mass index. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures and quality criteria follow the Statistical Analysis Plan (SAP).
Change from Baseline in Waist Circumference (cm) | Baseline, and 12 months post-surgery
  Waist circumference is measured in cm at the midpoint between the lowest rib and the iliac crest. Higher values indicate greater central adiposity. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurements follow standardized anthropometric procedures and the Statistical Analysis Plan.
Change from Baseline in Handgrip Strength (kg) | Baseline, and 12 months post-surgery
  Handgrip strength is assessed with a calibrated dynamometer; the best of repeated maximal trials is recorded in kg. Higher values indicate greater muscle strength. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures and test standardization follow the Statistical Analysis Plan.
Change from Baseline in Knee Extension Strength (Nm) | Baseline, and 12 months post-surgery
  Maximal voluntary knee extension strength is measured using a standardized dynamometer and recorded in Newton-meters (Nm). Higher values indicate greater quadriceps strength. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement procedures and calibration follow the device manual and the Statistical Analysis Plan.
Change from Baseline in Countermovement Jump Height (cm) | Baseline, and 12 months post-surgery
  Countermovement jump (CMJ) height is measured using a force platform or validated optical system and reported in cm. Higher values indicate better lower-body power. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Testing follows standardized procedures and the Statistical Analysis Plan.
Change from Baseline in Aortic Systolic Blood Pressure (SBPao, mmHg) | Baseline, 1-2 months, and 12 months post-surgery
  Aortic systolic pressure (SBPao) measured by Arteriograph under standardized resting conditions (10-12 h fast, no vigorous physical activity in prior 24 h, supine, thermoneutral room). Unit mmHg; higher value = higher SBPao. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures and quality criteria follow the device manual and the Statistical Analysis Plan.
Change from Baseline in Aortic Diastolic Blood Pressure (DBPao, mmHg) | Baseline, 1-2 months, and 12 months post-surgery
  Aortic diastolic pressure (DBPao) by Arteriograph in standardized rest (as above). mmHg; higher value = higher DBPao. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures follow the device manual and the Statistical Analysis Plan.
Change from Baseline in Aortic Pulse Pressure (PPao, mmHg) | Baseline, 1-2 months, and 12 months post-surgery
  Central pulse pressure = SBPao - DBPao by Arteriograph in standardized rest (as above). mmHg; higher = greater central pulsatility. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Device procedures follow the manual and the Statistical Analysis Plan.
Change from Baseline in Reflection Time (RT, ms) | Baseline, 1-2 months, and 12 months post-surgery
  Reflection time measured by Arteriograph in standardized rest (as above). ms; shorter RT = faster wave return. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement and quality criteria follow the device manual and the Statistical Analysis Plan.
Change from Baseline in Microvascular Perfusion (PU) | Baseline, 1-2 months, and 12 months post-surgery
  Resting cutaneous microvascular perfusion measured at the forearm using Laser Doppler under standardized resting conditions (10-12 h fast, no vigorous physical activity in prior 24 h, supine, thermoneutral). Perfusion units (PU); higher = higher resting microvascular flow. TThe outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement and quality criteria follow the Statistical Analysis Plan.
Change from Baseline in Endothelium-Dependent Vasodilation (Laser Doppler, %) | Baseline, 1-2 months, and 12 months post-surgery
  Endothelium-dependent vasodilatory response measured at the forearm using Laser Doppler during standardized forearm occlusion to induce a controlled ischemic stimulus under resting conditions (as above). % change from baseline; higher = better endothelial function. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Procedures follow the Statistical Analysis Plan.
Change from Baseline in Post-Occlusive Reactive Hyperemia (PORH, %) | Baseline, 1-2 months, and 12 months post-surgery
  Post-occlusive reactive hyperemia measured at the forearm with Laser Doppler under standardized rest (as above). % increase; higher = better microvascular reactivity. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Protocol and analysis follow the Statistical Analysis Plan.
Change from Baseline in Resting Near-Infrared Spectroscopy (NIRS) Tissue Oxygen Saturation (StO2, %) | Baseline, 1-2 months and 12 months post-surgery
  Near-Infrared Spectroscopy (NIRS)-derived quadriceps StO2 at rest under standardized conditions (10-12 h fast, no vigorous PA in prior 24 h, supine, thermoneutral). %; higher = higher oxygenation. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Probe placement/quality criteria per Statistical Analysis Plan.
Change from Baseline in Minimum Near-Infrared Spectroscopy (NIRS) Tissue Oxygen Saturation (StO2) During Exercise (%) | Baseline, and 12 months post-surgery
  Lowest quadriceps StO2 during a standardized cycle ergometer test (pre-test: 10-12 h fast, no vigorous PA in prior 24 h). %; lower value = deeper deoxygenation. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Exercise protocol and artifact handling per Statistical Analysis Plan.
Change from Baseline in Near-Infrared Spectroscopy (NIRS) Tissue Oxygen Saturation (StO2) Recovery Slope After Exercise (%/s) | Baseline, and 12 months post-surgery
  Slope of StO2 increase immediately after exercise cessation in standardised protocol (same pre-test conditions). %/s; steeper slope = faster microvascular reoxygenation. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Processing/quality criteria per Statistical Analysis Plan.
Change from Baseline in Near-Infrared Spectroscopy (NIRS) Total Hemoglobin (tHb, au) | Baseline, 1-2 months, and 12 months post-surgery
  NIRS-derived tHb signal (rest and/or during exercise, per protocol). Arbitrary units; marker of local microvascular blood volume. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Signal processing and artifact rejection per Statistical Analysis Plan.
Change from Baseline in Peak Oxygen Uptake (VO2peak, mL/kg/min) | Baseline, and 12 month post-surgery
  Peak oxygen uptake will be determined during a submaximal cycling test on an electronically braked ergometer with breath-by-breath indirect calorimetry under standardized pre-test conditions (10-12 h fast; avoid vigorous physical activity in the prior 24 h). VO2peak is expressed as mL/kg/min; higher values indicate better aerobic capacity. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Test protocol, stage structure, termination criteria and data processing follow the Statistical Analysis Plan.
Change from Baseline in Resting Fat Oxidation Rate (g/min) | Baseline, 1-2 month and 12 months post-surgery
  Resting whole-body fat oxidation will be assessed by indirect calorimetry (hood) before exercise under standardized conditions (10-12 h fast; no vigorous physical activity in the prior 24 h, supine/seated, thermoneutral). Rate is expressed as g/min (calculated from VO2 and VCO2 using standard stoichiometric equations); higher values indicate higher fat oxidation at rest. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Measurement details and calculations follow the Statistical Analysis Plan.
Change from Baseline in Maximal Fat Oxidation Rate (MFO, g/min) | Baseline, 1-2 month and 12 months post-surgery
  Maximal fat oxidation rate (MFO) will be derived from indirect calorimetry during the cycling fat oxidation assessment (per protocol), expressed in g/min; higher values indicate greater maximal fat oxidation capacity. Pre-test conditions: 10-12 h fast and no vigorous physical activity during the prior 24 h. The outcome is the change from baseline to the specified follow-up (follow-up - baseline). Stage definition, steady-state criteria, and computational details (e.g., selection of the maximal value) follow the Statistical Analysis Plan.
Change from Baseline in Rate of Torque Development (Nm/s) | Baseline to 1-2 months and 12 months post surgery.
  Rate of torque development (RTD) is derived from the isometric elbow flexion force-time signal recorded concurrently with electromyography (EMG) during the StartReact test under standardised pre-test conditions (10-12 h fast; no vigorous physical activity within 24 h; thermoneutral room, seated position). Force values for maximum voluntary contraction (MVC, N) are converted to torque (N·m) using each participant's individual lever arm distance measured from the humeroradial joint space to the centre of the strain gauge at the wrist. RTD is calculated as the slope of the force-time curve over the early contraction phase (first 50 ms) and expressed as torque rate (Nm/s). The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, and analysis are defined in the Statistical Analysis Plan.
Change from Baseline in Voluntary Electromyography Amplitude (µV) | Baseline to 1-2 months and 12 months post surgery.
  Voluntary electromyography (EMG) amplitude over the initial 50 ms window recorded during the StartReact test under the same standardised pre-test conditions. EMG amplitude is expressed in microvolts (µV). The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, and analysis are defined in the Statistical Analysis Plan.
Change from Baseline in Short Interval Intracortical Inhibition (SICI) [% of comparator MEP amplitude] | Baseline to 1-2 months and 12 months post surgery
  Short interval intracortical inhibition (SICI) will be assessed using a paired pulse transcranial magnetic stimulation (TMS) paradigm in which a subthreshold conditioning stimulus precedes a suprathreshold test stimulus at a short interstimulus interval (typically 2-5 ms). Electromyography (EMG) from the biceps brachii is recorded under standardised pre-test conditions (10-12 h fast; no vigorous physical activity within 24 h; thermoneutral room; consistent coil positioning). The analysis variable for this outcome is the percentage inhibition of the test pulse motor evoked potential (MEP) relative to the MEP amplitude elicited using the single pulse condition (comparator MEP). Lower values indicate stronger intracortical inhibition. The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, stimulus parameters, trial rejection rules, and averaging procedures follow the Statistical Analysis Plan.
Change from Baseline in Long Interval Intracortical Inhibition (LICI) [% of comparator MEP amplitude] | Baseline to 1-2 months and 12 months post surgery
  Long interval intracortical inhibition (LICI) will be assessed using a paired pulse TMS paradigm in which a suprathreshold conditioning pulse precedes a suprathreshold test pulse at a long interstimulus interval (typically 50-200 ms). Electromyography (EMG) from the biceps brachii is recorded under the same standardised pre-test conditions used for SICI assessment. The analysis variable for this outcome is the percentage inhibition of the test pulse motor evoked potential (MEP) relative to the MEP amplitude elicited using the single pulse condition (comparator MEP). Lower values indicate stronger intracortical inhibition. The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, stimulus parameters, trial rejection rules, and averaging procedures follow the Statistical Analysis Plan.
Change from Baseline in Intra Cortical Facilitation (ICF) [% of comparator MEP amplitude] | Baseline to 1-2 months and 12 months post surgery
  Intra-cortical facilitation (ICF) will be assessed using a paired pulse transcranial magnetic stimulation (TMS) paradigm in which a subthreshold conditioning stimulus precedes a suprathreshold test stimulus at an interstimulus interval that facilitates corticospinal output (typically 8-20 ms). Electromyography (EMG) from the biceps brachii is recorded under standardised pre-test conditions (10-12 h fast; no vigorous physical activity within 24 h; thermoneutral room; consistent coil positioning). The analysis variable for this outcome is the percentage facilitation of the test pulse motor evoked potential (MEP) relative to the MEP amplitude elicited using the single pulse condition (comparator MEP). Higher values indicate stronger intracortical facilitation. The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, stimulus parameters, trial rejection rules, and averaging procedures follow the Statistical Analysis Plan.
Change from Baseline in StartleTMS Response [% of comparator MEP amplitude] | Baseline to 1-2 months and 12 months post surgery
  StartleTMS will be assessed using a paired single pulse transcranial magnetic stimulation (TMS) protocol in which a loud acoustic stimulus precedes the TMS pulse, eliciting startle related facilitation of corticospinal output. Electromyography (EMG) from the biceps brachii is recorded under standardised pre-test conditions (10-12 h fast; no vigorous physical activity within 24 h; thermoneutral room; consistent coil positioning). The analysis variable for this outcome is the percentage change in motor evoked potential (MEP) amplitude under the StartleTMS condition relative to the MEP amplitude elicited during the single pulse comparator condition. Higher values indicate stronger startle related facilitation of corticospinal excitability. The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, stimulus parameters, trial rejection rules, and averaging procedures follow the Statistical Analysis Plan.
Change from Baseline in Silent Period Duration Normalised to MEP [ms/MEP] | Baseline to 1-2 months and 12 months post surgery
  The silent period (SP) will be derived from the interruption in voluntary electromyography (EMG) activity following a suprathreshold single pulse transcranial magnetic stimulation (TMS) stimulus delivered during the stimulus-response curve test. SP duration is first measured in milliseconds (ms) from the motor evoked potential (MEP) onset to the resumption of voluntary EMG activity and then normalised to MEP amplitude (expressed as ms/MEP) for between timepoint comparisons. The outcome is the change from baseline to follow up (follow up - baseline). Condition, quality criteria, detection thresholds, stimulus parameters, and averaging procedures follow the Statistical Analysis Plan.
Hormonal Regulation of Adipose Tissue Health and Cellular Function | Tissue samples will be collected during surgery, likely between March 2026 to December 2027, followed by Adipoid development within a week of collection. Exposure experiments of the Adipoids will use time frames from onset up to 48 hours.
  This is an exploratory laboratory outcome. Adipose Organoids (Adipoids) will be exposed to a variety of hormonal environments created with either pure hormone substances or condition media supplemented with pre- and postmenopausal sera. Readouts include change in Adipoid cellular content (cell count, number of cells/ml). Additional exploratory variables will be collected and may be analyzed; these are listed as exploratory Other Prespecified Outcomes, including lipid uptake, reaction on inflammatory stimuli, gene expression or secretome, in the Statistical Analysis Plan.

CONTACTS AND LOCATIONS:
Overall Officials: Eija K Laakkonen, Associate Professor, Principal Investigator — University of Jyvaskyla

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy regulations and GDPR compliance. Summary results will be published in peer-reviewed journals and presented at scientific conferences. The study protocol will be published as an open-access article. Supporting documents such as the statistical analysis plan, analytic code, informed consent form (blank version), questionnaires, and standard operating procedures (SOPs) will be available upon reasonable request. Aggregated, anonymised data may be shared upon reasonable request for research purposes, subject to ethical approval and data-sharing agreements.

REFERENCES:
- See also: Home page of the HoCa study — https://www.jyu.fi/en/projects/hormonal-regulation-of-cardiometabolic-health-hoca